CLINICAL TRIAL: NCT00538122
Title: Evaluating the Risks of Arrhythmia and Sudden Death Associated With Antipsychotic Drugs by Assessing the T Wave Abnormalities in the Holter Electrocardiogram
Brief Title: Changes in Heart Rhythms Associated With Antipsychotic Drug Treatment
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Herbert Meltzer, M.D., Vanderbilt University Medical Center
Other Study IDs: 070591
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
Keywords: schizophrenia; schizoaffective disorder; bipolar disorder; antipsychotic drug treatment; safety; arrythmias
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thioridazine Group: Patients must have been treated with (Mellaril) thioridazine at least three months at time of enrollment.
  Interventions: Device: 24 Holter Monitor Recording

INTERVENTIONS:
Device: 24 Holter Monitor Recording — All subjects will be fitted with a device to obtain 24-hour Holter EKG continuous recordings of bipolar leads C5C5R. They will also receive a standard 12-lead EKG recording prior to the placement of the Holter device. The subjects will be asked to keep a diary during the course of the 24 hours to record information such as wake and sleep times and symptoms such as shortness of breath, heart palpitations, lightheadedness, etc.
  From each recording, 12 sets of 10 consecutive QRS epochs, plus QRS samplings obtained during sleep will be analyzed by a cardiologist blind to the medication status of subjects.

SUMMARY:
This study is being done to look at the electrical activity of the heart. This study will help decide whether taking recordings for a 24-hour period gives more useful information than recording it for a few seconds in a doctor's office. The study will compare 24 hour electrocardiogram (ECG) results of patients taking thioridazine (Mellaril) to those of other patients taking different medications that took part in another study.

DETAILED DESCRIPTION:
The objective of the study is to assess the Tpe and QTc measures in 24 hr Holter echocardiograms in patients treated with atypical antipsychotic drgs (APDs). The primary comparisons of interest are olanzapine (no QTc prolongation) to ziprasidone (QTc prolongation) and thioridazine (QTc prolongation) as well as ziprasidone (possibly low TdP risk) to thioridazine (TdP risk). Secondary comparisons will be among all APDs available. In a previously approved study, conventional 24 hr Holter electrocardiograms were recorded from a total of 78 subjects during the course of treatment with psychotropic medications and without medication (in the case of normals and unmedicated patients). These recordings will be analyzed to yield Tpe, QTc and heart rate, and other measures. Data from additional patients is needed, therefore this study will include only patients currently treated with Mellaril (thioridazine), Risperdal (risperidone) and Seroquel (quetiapine).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be male or female, age 18-65

  * Patients must have a definitive diagnosis by DSM-IV criteria of schizophrenia, bipolar or schizoaffective disorder.
  * Patients can be receiving inpatient or outpatient treatment at time of enrollment.
  * Patients must have been treated with (Mellaril) thioridazine, (Risperdal) risperidone or (Seroquel) quetiapine at least three months at time of enrollment.
  * Patients must be able to provide written informed consent

Exclusion Criteria:

* Patients with a primary diagnosis other than schizophrenia, schizoaffective or bipolar disorder

  * Patients who are currently taking other medications that have been shown to prolong the QTC, including tricyclic antidepressants, fluoroquinolones or antiarrythmics.
  * Patients unable to provide written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed wtih schizophrenia, bipolar or schizoaffective disorder
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Meltzer, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Psychiatric Hospital, Nashville, Tennessee, United States